CLINICAL TRIAL: NCT06941337
Title: HEALTHYSTEPS + PLAYREADVIP EFFECTS ON PARENTING AND CHILD DEVELOPMENT: A RANDOMIZED IMPLEMENTATION EFFECTIVENESS TRIAL
Brief Title: HealthySteps + PlayReadVIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-01988; 1R01MD018597 (NIH)
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Families With Infants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthySteps + PlayReadVIP (Experimental): Families (parent-child dyads) randomized to receive HealthySteps (HS), which provides parenting support, plus PlayReadVIP, which promotes relational health through video coaching.
  Interventions: Behavioral: HealthySteps (HS); Behavioral: PlayReadVIP
- Standard HealthySteps (Active Comparator): Families (parent-child dyads) randomized to receive HealthySteps (HS), which provides parenting support, only.
  Interventions: Behavioral: HealthySteps (HS)

INTERVENTIONS:
Behavioral: HealthySteps (HS) — Evidence-based program that focuses on addressing Adverse Childhood Experiences (ACEs) and family stressors. The program provides parenting guidance, mental health support, and care coordination. The program is delivered during well-child visits by an HS specialist.
Behavioral: PlayReadVIP — Evidence-based program that promotes Positive Childhood Experiences (PCEs) and strengthens parent-child interactions. The program involves recording and reviewing videos of parents engaging with their child to provide feedback and encourage positive practices. Families receive toys, books, and guides to extend activities at home.
  Arms: HealthySteps + PlayReadVIP

SUMMARY:
This study aims to investigate the effectiveness and implementation outcomes for the integration of two evidence-based practices and interventions (EBPIs) within pediatric primary care settings: HealthySteps (HS), which provides parenting support, and PlayReadVIP, which promotes relational health through video coaching. Families will be randomized to receive either the integrated HS + PlayReadVIP model or traditional HS, and investigators will examine impacts on parenting, parent-child relationships, and child development, as well as feasibility, acceptability, and appropriateness of the integrated intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parent is a biological parent or legal guardian and at least 18 years of age
* Infants must be ≤6 months old at the time of enrollment.
* Parents/guardians must speak either English or Spanish to ensure they can fully engage with the intervention and assessments.
* Families must be identified as Tier 3 HealthySteps participants, indicating higher levels of need based on clinic screening for factors such as:Adverse Childhood Experiences (ACEs) and parenting challenges or vulnerabilities.
* Parent is able to willing to provide consent for their own and their child's participation.

Exclusion Criteria:

* Non-singleton child
* Parent is unable to provide consent
* Parent does not speak English or Spanish, as study materials (e.g., questionnaires) are available in those languages
* Parent has a severe medical or psychiatric impairment (e.g., intellectual disability, psychosis) that would interfere with study participation
* Parent has plans to discontinue care at NYU Langone Health - Sunset Park Family Health Centers

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Adult-Child Relationship Scale Score | Month 12
  13-item assessment of parent-child relationship quality. Each item is rated on a Likert 5 scale from 1 (definitely not) to 5 (definitely). The total score is the average of item responses and ranges from 1-5; higher scores indicate a stronger and more positive relationship between the child and parent.
Adult-Child Relationship Scale Score | Month 24
  13-item assessment of parent-child relationship quality. Each item is rated on a Likert 5 scale from 1 (definitely not) to 5 (definitely). The total score is the average of item responses and ranges from 1-5; higher scores indicate a stronger and more positive relationship between the child and parent.
Stimulation Questionnaire (StimQ) Core: Reading, Teaching, Verbal Responsivity Score | Month 12
  The StimQ is a parent-report measure of the cognitive home environment, designed to assess the level of cognitive stimulation children receive at home. Items include dichotomous (yes or no) and Likert-style responses ranging from 0-4. The total score is the sum of item responses and ranges from 0 to 43; higher scores are correlated with better parental behavior.
Stimulation Questionnaire (StimQ) Core: Reading, Teaching, Verbal Responsivity Score | Month 24
  The StimQ is a parent-report measure of the cognitive home environment, designed to assess the level of cognitive stimulation children receive at home. Items include dichotomous (yes or no) and Likert-style responses ranging from 0-4. The total score is the sum of item responses and ranges from 0 to 43; higher scores are correlated with better parental behavior.
Infant Behavior Questionnaire Score | Month 12
  36-item parent-report questionnaire used to measure the temperament of an infant (3-12 months old). Each item is rated on a scale from 1 (never) to 7 (always); the total score is the average of responses and ranges from 1-7; higher scores indicating greater frequency of behaviors.
Brief Infant Toddler Social-Emotional Assessment (BITSEA) Score: Competence | Month 12
  BITSEA measures socioemotional development in toddlerhood. 11 of the items cover competence. Each item is rated on a scale from 0-2. The total BITSEA Competence Score is the sum of responses and ranges from 0-22; higher scores indicate greater functioning.
Brief Infant Toddler Social-Emotional Assessment (BITSEA) Score: Problems | Month 12
  BITSEA measures socioemotional development in toddlerhood. 31 of the items cover problems. Each item is rated on a scale from 0-2. The total BITSEA Problems Score is the sum of responses and ranges from 0-62; higher scores indicate poorer functioning.
Child Behavior Checklist Score | Month 24
  100-item questionnaire identifying problem behavior in children. Each item is rated on a scale from 0 (absent) to 2 (often occurs). The raw score is the sum of responses and is transformed into a final t-score ranging from 0-100 with a mean of 50 and standard deviation of 10. T-scores below 60 indicate non-clinical symptoms; t-scores between 60 and 64 indicate that the child is at risk for problem behaviors; and t-scores above 65 indicate clinical symptoms.

SECONDARY OUTCOMES:
Edinburgh Depression Scale (EPDS) Score | Baseline
  10-item screening tool used to assess symptoms of depression in pregnant and postpartum women. The total score is determined by adding together the scores for each of the 10 items and ranges from 0-30; higher scores indicate greater severity of depression.
Edinburgh Depression Scale (EPDS) Score | Month 12
  10-item screening tool used to assess symptoms of depression in pregnant and postpartum women. The total score is determined by adding together the scores for each of the 10 items and ranges from 0-30; higher scores indicate greater severity of depression.
Edinburgh Depression Scale (EPDS) Score | Month 24
  10-item screening tool used to assess symptoms of depression in pregnant and postpartum women. The total score is determined by adding together the scores for each of the 10 items and ranges from 0-30; higher scores indicate greater severity of depression.
Perceived Stress Scale (PSS) Score | Baseline
  10-item assessment of stress over the past month. Each item is rated on a scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0-40; higher scores indicate more severe stress.
Perceived Stress Scale (PSS) Score | Month 12
  10-item assessment of stress over the past month. Each item is rated on a scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0-40; higher scores indicate more severe stress.
Perceived Stress Scale (PSS) Score | Month 24
  10-item assessment of stress over the past month. Each item is rated on a scale from 0 (never) to 4 (very often). The total score is the sum of responses and ranges from 0-40; higher scores indicate more severe stress.
Parenting Self-Agency Measure | Baseline
  5-item assessment of thoughts and feelings about being a parent. Each item is rated on a scale from 1 (almost never or never) to 5 (almost always or always). The total score ranges from 5-25; higher scores indicate greater parenting self-agency.
Parenting Self-Agency Measure | Month 12
  5-item assessment of thoughts and feelings about being a parent. Each item is rated on a scale from 1 (almost never or never) to 5 (almost always or always). The total score ranges from 5-25; higher scores indicate greater parenting self-agency.
Parenting Self-Agency Measure | Month 24
  5-item assessment of thoughts and feelings about being a parent. Each item is rated on a scale from 1 (almost never or never) to 5 (almost always or always). The total score ranges from 5-25; higher scores indicate greater parenting self-agency.
Patient-Reported Outcomes Measurement Information System (PROMIS): General Life Satisfaction Scale Score | Baseline
  5-item questionnaire of life satisfaction. Responses are scored on a Likert scale and then converted to a T-score with a mean of 50 and a standard deviation of 10, where higher scores indicate greater satisfaction.
PROMIS: General Life Satisfaction Scale Score | Month 12
  5-item questionnaire of life satisfaction. Responses are scored on a Likert scale and then converted to a T-score with a mean of 50 and a standard deviation of 10, where higher scores indicate greater satisfaction.
PROMIS: General Life Satisfaction Scale Score | Month 24
  5-item questionnaire of life satisfaction. Responses are scored on a Likert scale and then converted to a T-score with a mean of 50 and a standard deviation of 10, where higher scores indicate greater satisfaction.
Dyadic Adjustment Scale Score | Baseline
  32-item assessment of relationship quality of intact couples. Each item is rated on a scale; the total score is the sum of responses. Scores range from 0 to 151, with higher scores indicating greater relationship satisfaction and lower scores suggesting more distress.
Dyadic Adjustment Scale Score | Month 12
  32-item assessment of relationship quality of intact couples. Each item is rated on a scale; the total score is the sum of responses. Scores range from 0 to 151, with higher scores indicating greater relationship satisfaction and lower scores suggesting more distress.
Dyadic Adjustment Scale Score | Month 24
  32-item assessment of relationship quality of intact couples. Each item is rated on a scale; the total score is the sum of responses. Scores range from 0 to 151, with higher scores indicating greater relationship satisfaction and lower scores suggesting more distress.
Socolar Discipline Survey Score | Month 12
  34-item questionnaire assessing how a parent handles their problems with their children's behavior over the past 3 months. Each item is rated on a scale from 1 (never) to 6 (always). The total score is the sum of responses and ranges from 34 to 204; higher scores indicate greater frequency of harsher discipline.
Socolar Discipline Survey Score | Month 24
  34-item questionnaire assessing how a parent handles their problems with their children's behavior over the past 3 months. Each item is rated on a scale from 1 (never) to 6 (always). The total score is the sum of responses and ranges from 34 to 204; higher scores indicate greater frequency of harsher discipline.
Early Social Communication Scale (ESCS) Score | Month 12
  The ESCS is a videotaped, structured observation measure designed to assess nonverbal communication skills in children. Frequency scores for initiation of joint attention (IJA) are derived from behavioral observations during a series of tasks. IJA score ranges from 0 to 100 where a higher value indicates greater initiation of joint attention.
Early Social Communication Scale (ESCS) Score | Month 24
  The ESCS is a videotaped, structured observation measure designed to assess nonverbal communication skills in children. Frequency scores for initiation of joint attention (IJA) are derived from behavioral observations during a series of tasks. IJA score ranges from 0 to 100 where a higher value indicates greater initiation of joint attention.
MacArthur-Bates Communicative Development Inventory (CDI) Score | Month 12
  Parent report instrument that measures early language development, including productive vocabulary. Parents mark each example of words that their child says. The total score is the total number of words marked.
MacArthur-Bates Communicative Development Inventory (CDI) Score | Month 24
  Parent report instrument that measures early language development, including productive vocabulary. Parents mark each example of words that their child says. The total score is the total number of words marked.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Caitlin, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: caitlin.canfield@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to caitlin.canfield@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.